CLINICAL TRIAL: NCT01277172
Title: Comparative,Randomized,Double Blind Study to Evaluate Biologic Effect and Safety of PBO-326 (Rituximab), Associated to CHOP-14 Compared With Mabthera (Rituximab) Associated to CHOP-14 in B Cells CD20+ Diffuse Non-Hodgkin Lymphoma Patients
Brief Title: TREatment of degeNerative and Neoplastic Diseases With Rituximab
Acronym: TREND
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Probiomed S.A. de C.V. (Industry)
Responsible Party: Jorge Revilla Beltri, MD., Probiomed, S.A. de C.V.
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO-1908; PRO1908TREND (Other: PRO1908TREND012011)
Record Dates: First submitted 2011-01-08; First posted 2011-01-14 (Estimated); Last update posted 2011-01-14 (Estimated); Status verified 2011-01

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: DLBCL; pharmacokinetics; pharmacodynamics; Rituximab; LymphomaLymphoma; Non-HodgkinLymphoma; B-CellLymphoma; Large B-Cell; Disorders Lymphatic Diseases; Immunoproliferative Disorders; Antineoplastic Agents; Adverse Effects
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Immunoproliferative Disorders | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 / PBO-326 (Experimental): This group will be treated three cycles with PBO-326, after the third cycle the patients will receive Mabthera for another three cycles.
  Interventions: Biological: Rituximab
- Group 2 / Mabthera (Active Comparator): This group will be treated three cycles with Mabthera, after the third cycle the patients will receive PBO-326 for another three cycles.
  Interventions: Biological: Rituximab
- Group 3 / PBO-326 (Experimental): This group will be treated six cycles with PBO-326
  Interventions: Biological: Rituximab
- Group 4 / Mabthera (Active Comparator): This group will be treated six cycles with Mabthera
  Interventions: Biological: Rituximab

INTERVENTIONS:
Biological: Rituximab — 375 mg/m2 IV every 2 weeks for 6 cycles
  Other Names: Monoclonal Antibody against CD20
  Arms: Group 1 / PBO-326
Biological: Rituximab — 375 mg/m2 IV every 2 weeks for 6 cycles
  Other Names: Monoclonal Antibody against CD20
  Arms: Group 2 / Mabthera
Biological: Rituximab — 375 mg/m2 IV every 2 weeks for 6 cycles
  Other Names: Monoclonal Antibody against CD20
  Arms: Group 3 / PBO-326
Biological: Rituximab — 375 mg/m2 IV every 14 days for 6 cycles
  Other Names: Monoclonal antibody against CD20
  Arms: Group 4 / Mabthera

SUMMARY:
This is a prospective international, multi-center, randomized, double-blind controlled study designed to assess and compare the pharmacokinetics, pharmacodynamics and the safety of PBO-326 (Rituximab) and Mabthera (Rituximab) in combination with CHOP in previously untreated patients with diffuse B cells Non Hodgkin lymphoma.

DETAILED DESCRIPTION:
At present R-CHOP (Rituximab plus Cyclofosfamide, Doxorrubicine, Vincristine and Prednisone) has became standard of care of patients with B cells Non Hodgkin Lymphoma CD20+.

Study will perform pharmacodynamic (PD) and pharmacokinetic (PK) measurment of a novel Rituximab in comparison with Mabthera and evaluates safety both metabolic as well immunologic.

Study protocolo is designed to provide data on impact of treatment interchange of both study drugs (PBO-326 and Mabthera).

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed subjects with a confirmed pathologic diagnosis of diffuse large B cell non-Hodgkin's lymphoma (DLBCL) based on the 2008 World Health Organization classification.
2. CD20+ lymphoma cells at screening.
3. > 18 years of age at screening.
4. Ann Arbor Stages I-IV at screening.
5. Any IPI score at screening.
6. Easten Cooperative Oncology Group (ECOG) performance status (0-2) or Karnofsky scale > 60 at screening.
7. Left ventricular ejection fraction > 50%.
8. Willing and able to provide written informed consent prior to performing study procedures.
9. Women of childbearing potential must use effective contraceptive methods starting from screening and until 12 months following the last infusion.

Exclusion Criteria:

1. Hodgkin lymphoma.
2. Any lymphoma other than CD20+ Diffuse Large B Cell Lymphoma (DLBCL).
3. Immunodeficiency syndrome or Human immunodeficiency virus (HIV) seropositivity .
4. Active uncontrolled infection (viral, bacterial or fungal infection) requiring systemic therapy at screening and/or at baseline visit.
5. Function Liver tests >2 x upper normal values.
6. Positive Hepatitis B surface antigen or antibodies to Hepatitis C.
7. Any other serious active disease or co-morbid medical condition.
8. Subjects who, according to the investigator, are likely to be non-compliant or uncooperative during the study.
9. Pregnant or breast-feeding women or women that intend to get pregnant during study or within 12 months following the last infusion.
10. Treatment with any investigational drug within 90 days before day 1 of study treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-09 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Basal and final serum CD 20 levels comparison. | Every 14 days for the duration of treatment
  Primary outcome is the depletion of CD20+ B cells. This will be measured every 14 days and comparison will be made basal levels versus visit 2, visit 3, visit 4, visit 5, visit 6, visit 7 and visit 8.

SECONDARY OUTCOMES:
Comparison of safety of PBO-326 versus Mabthera | Every 14 days measurements
  Adverse events will be observed and recorded in relation to acute infusion events (number of cases and severity of hypotension, hipertension, headache, and all cardiovascular events previously reported by Mabthera) as well as long term effects over key hematological cells (number of cases and severity of neutropenia, trombocytopenia, leucopenia) per visit.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Revilla Beltri, MD, Study Director — Probiomed S.A. de C.V.
Locations (1):
- INCan, México, D.f., Mexico